CLINICAL TRIAL: NCT00000688
Title: A Randomized, Controlled Study of Intravenous Ganciclovir Therapy for Peripheral Cytomegalovirus Retinitis in Patients With AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Purpose: Treatment
Other Study IDs: ACTG 071; RS-21592; ICM 1697
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1990-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Injections, Intravenous; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To provide information about the usefulness and safety of giving injections of ganciclovir (DHPG) for treating peripheral cytomegalovirus (CMV) retinitis.

CMV retinitis is an important sight-threatening opportunistic infection which affects 1 to 2 out of every 10 patients with AIDS. Results from an earlier study suggest that about 80 percent of patients with CMV retinitis will be helped by receiving intravenous doses of DHPG.

DETAILED DESCRIPTION:
CMV retinitis is an important sight-threatening opportunistic infection which affects 1 to 2 out of every 10 patients with AIDS. Results from an earlier study suggest that about 80 percent of patients with CMV retinitis will be helped by receiving intravenous doses of DHPG.

Patients are randomly placed in one of two treatment groups. In one group, patients receive DHPG twice a day, intravenously, for 14 days, followed by a daily dose for 14 weeks. Patients in the other group (the delayed-treatment group) do not receive immediate treatment with DHPG. Patients in both groups have regular ophthalmologic (eye) evaluations with retinal photographs to see if the retinitis is getting worse. Patients in the delayed treatment group receive DHPG if this occurs.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT) for patients in delayed treatment group and not receiving ganciclovir.
* Didanosine (ddI) may be continued or initiated in any patient during the study.
* Topical acyclovir.
* Topical ophthalmics.
* Aerosolized pentamidine.

Patients must have:

* AIDS as defined by the CDC criteria or have had confirmation of HIV infection by ELISA, p24 antigen assay, or culture of HIV.
* Retinal lesions greater than 1500 microns from edge of optic disc outside major temporal vascular arcades, and greater than 3000 microns from fovea.
* Understanding of study provisions, and willingness to sign informed consent form approved by the appropriate Institutional Review Board and Syntex.
* Life expectancy of at least 4 months.

Exclusion Criteria

Co-existing Condition:

Patients with ocular conditions requiring immediate surgical correction are excluded.

Concurrent Medication:

Excluded during first 4 weeks of ganciclovir treatment:

Zidovudine (AZT).

Excluded:

Other investigational drugs and antimetabolites, alkylating agents, nucleoside analogs (topical ophthalmics are permitted), acyclovir, interferon, foscarnet (non-nucleoside pyrophosphate analog), cytomegalovirus (CMV) hyperimmune globulin, and cytokines.

Patients with the following are excluded:

* Immediately sight-threatening retinitis (= or < 1500 microns from edge of optic disc, or inside major temporal vascular arcades, or = or < 3000 microns from the fovea).
* Ocular media opacities (corneal, lenticular, or vitreal) preventing ophthalmologic and photographic retinal assessment.
* Demonstrated hypersensitivity to acyclovir.

Prior Medication:

Excluded:

- Previous treatment with anti-cytomegalovirus therapy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180
Dates: Primary Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spector SA, Study Chair; Jabs D, Study Chair
Locations (22):
- United States (22):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Mount Zion Med Ctr, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Pacific Presbyterian, San Francisco, California
  - Mills Hosp, San Mateo, California
  - Stanford Univ School of Medicine, Stanford, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Henry Ford Hosp, Detroit, Michigan
  - Univ of Minnesota, Minneapolis, Minnesota
  - Kansas City Veterans Administration Med Ctr, Kansas City, Missouri
  - Washington Univ Med Ctr, St Louis, Missouri
  - Univ of New Mexico Hlth Sciences Ctr / Dept of Med, Albuquerque, New Mexico
  - New York Univ Med Ctr / Dept of Environmental Med, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Plaza Med Ctr, Houston, Texas
  - Infectious Diseases Association of Houston / Methodist Hosp, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia

REFERENCES:
- [Background] Spector SA, Weingeist T, Pollard RB, Dieterich DT, Samo T, Benson CA, Busch DF, Freeman WR, Montague P, Kaplan HJ, et al. A randomized, controlled study of intravenous ganciclovir therapy for cytomegalovirus peripheral retinitis in patients with AIDS. AIDS Clinical Trials Group and Cytomegalovirus Cooperative Study Group. J Infect Dis. 1993 Sep;168(3):557-63. doi: 10.1093/infdis/168.3.557. PMID 8394858